CLINICAL TRIAL: NCT01017679
Title: Phase II Multi-centre Randomized Controlled Study of Gefitinib 500mg Versus 250mg in Patients With NSCLC With Stable Disease After a Month Treatment of Gefitinib 250mg
Brief Title: Gefitinib 500mg Versus 250mg in Patients With NSCLC With Stable Disease After a Month Treatment of Gefitinib 250mg
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Wu Jieping Medical Foundation (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-JC-003
Record Dates: First submitted 2009-11-10; First posted 2009-11-20 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2012-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Oral Drug gefitinib(Iressa) 500 mg Everyday
  Interventions: Drug: Gefitinib 500mg/Gefitinib 250mg
- 2 (Active Comparator): Oral Drug gefitinib(Iressa) 250 mg Everyday
  Interventions: Drug: Gefitinib 500mg/Gefitinib 250mg

INTERVENTIONS:
Drug: Gefitinib 500mg/Gefitinib 250mg — Gefitinib 500mg or 250mg is Taken Orally everyday by Experimental and controlled Arms respectively
  Other Names: Iressa

SUMMARY:
This is a multi-center phase II randomized controlled study to assess the efficacy of Gefitinib 500mg in patients with IIIB/IV staged non-small cell lung cancer(NSCLC) with stable disease after a month treatment of 250mg Gefitinib by DCR,also PFS and OS.The side effect is evaluated as well.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed stage IIIB/IV lung cancer(exclude patients confirmed by sputum cytology)
2. received at least one chemotherapy regimen
3. with stable disease after a month treatment of gefitinib(CT scan)
4. the radiotherapy focus is not the measurable disease within 4 weeks.the patients received palliative therapy can be included.
5. Age >18 years, either sex
6. with a measurable disease(longest diameters >=10mm with Spiral computed tomography (CT)and >=20mm with conventional CT) at least according to RECIST Criteria
7. WHO performance status(PS)<= 2 ( Patients Whit PS=2 Should not get worsen within 2 weeks Before Included)
8. N>=1.5×109/L, Plt>=1.5×109/L,Hb>=10g/dL
9. ALP<2.5×ULN.If ALP>=2.5ULN, AST&ALT should <1.5ULN(without liver metastasis) or <5ULN(with liver metastasis).TBIL<=1.5ULN，AST&ALT<2.5ULN(without liver metastasis) or <5ULN (with liver metastasis).
10. Signed and dated informed consent before the start of specific protocol procedures.
11. recruiting and receiving treatment in 5 days after last CT scan
12. Patients able to taken oral drug

Exclusion Criteria:

1. Life expectancy <= 12 weeks.Patients with metastatic brain tumors without symptoms or had been treated can be included.
2. experience of Anti-EGFR(the epidermal growth factor receptor) Monoclonal Antibody or small molecular compounds therapy such as erlotinib or Cetuximab.
3. can not take drug orally, have active peptic ulcer,half upper gastrointestinal or have dyspepsia.
4. allergic to gefitinib
5. Prior exposure to drugs without approval from this research or other study drugs within 21days before the 1st day taken Gefitinib 500mg or 250mg.
6. Pregnant or breast-feeding women
7. Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.
8. Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except of cervical carcinoma in situ,basal cell carcinoma within 5 years prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2009-05; Primary Completion 2012-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Comparing the difference of Response rate(CR & PR) | 3 years

SECONDARY OUTCOMES:
Comparing the difference of PFS(Progression Free Survival)and OS(Overall Survival) in two arms | 3 and a half years

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer Center of Sun-Yat Sen University, Guangzhou, Guangdong, China